CLINICAL TRIAL: NCT03061149
Title: The Effects of Nerve and Tendon Gliding Exercises Combined With Low-level Laser or Ultrasound Therapy in Carpal Tunnel Syndrome
Brief Title: The Effectiveness of Physical Therapy Modalities in Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Małgorzata Eliks, Assistant, Poznan University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1029/08
Record Dates: First submitted 2017-02-14; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group with low-level laser treatment (Experimental): The group received low-level laser therapy (LLLT). The application of a GaAlAs infrared laser with a pencil probe (BTL 5000 Combi, United Kingdom; at 830 nm, 9J/cm2 per point, power output of 100 mW, beam diameter of 5 mm) was performed at five points along the median nerve on the palmar side of the wrist 7. The time of exposure was 10 minutes (2 minutes per point). Both the patient and the therapist wore protective glasses during every session.A total of 10 therapeutic sessions were performed during a period of two weeks (five session times per week).
  Additionally, nerve and gliding exercises were administered.
  Interventions: Other: Low-level laser therapy
- Group with ultrasound treament (Active Comparator): The group underwent ultrasound treatment. Ultrasound treatment was administered at a frequency of 1 MHz, intensity of 1 W/cm2 ,pulsed mode duty cycle of 1:4 and with a handhold transducer of 5 cm2 (BTL 5000 Combi, UK). The time of application was 6 minutes over the area of the carpal tunnel. Aquasonic gel was used as a couplant. A total of 10 therapeutic sessions were performed during a period of two weeks (five session times per week). Additionally, nerve and gliding exercises were administered.
  Interventions: Other: Ultrasound treatment

INTERVENTIONS:
Other: Low-level laser therapy
  Arms: Group with low-level laser treatment
Other: Ultrasound treatment
  Arms: Group with ultrasound treament

SUMMARY:
Carpal tunnel syndrome is considered to be the most common entrapment neuropathy. Conservative treatment is recommended in the mild and moderate stage of CTS. The aim of this trial is to evaluate the effectiveness of physical therapy modalities in carpal tunnel syndrome.

DETAILED DESCRIPTION:
Conservative treatment is recommended in the mild and moderate stage of CTS and should involve splinting, steroid injections, oral steroids and ultrasounds .

However, the results of some research studies have showed the beneficial effect of photobiomodulation as well as nerve and tendon gliding exercises in non-operative treatment .

Patients were divided into two groups. The one group received low-level laser therapy (LLLT); the other group underwent ultrasound treatment. Additionally, nerve and gliding exercises were administered in both groups.

The purpose of this trial is to assess the therapeutic efficacy of ultrasound treatment and low-level laser therapy combined with nerve and tendon gliding exercises and to compare the two regimens.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of the mild or moderate stage of CTS, symptom duration for more than three months and general good health

Exclusion Criteria:

* advanced CTS, secondary CTS, any previous surgery in the upper limb, steroid injections and any physical therapy treatment within six months prior to the study, pregnancy, cervical radiculopathy, peripheral polyneuropathy or other neurological conditions

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2009-03-30 (Actual); Primary Completion 2014-02-15 (Actual); Study Completion 2016-11-12 (Actual)

PRIMARY OUTCOMES:
The measurement of hand grip strength in patients with carpal tunnel syndrome after physical therapy | 14 days
  The Jamar dynamometer (Sammons Preston, Canada) is used to assess hand grip strength; the mean score of three consecutive trials is accepted for each strength measurement. The result is expressed in kilogram [kg]. The evaluation is performed before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Małgorzata Zgorzalewicz-Stachowiak, PhD, Study Director — Poznan University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shooshtari SM, Badiee V, Taghizadeh SH, Nematollahi AH, Amanollahi AH, Grami MT. The effects of low level laser in clinical outcome and neurophysiological results of carpal tunnel syndrome. Electromyogr Clin Neurophysiol. 2008 Jun-Jul;48(5):229-31. PMID 18754533
- [Background] Rozmaryn LM, Dovelle S, Rothman ER, Gorman K, Olvey KM, Bartko JJ. Nerve and tendon gliding exercises and the conservative management of carpal tunnel syndrome. J Hand Ther. 1998 Jul-Sep;11(3):171-9. doi: 10.1016/s0894-1130(98)80035-5. PMID 9730093
- [Background] Ebenbichler GR, Resch KL, Nicolakis P, Wiesinger GF, Uhl F, Ghanem AH, Fialka V. Ultrasound treatment for treating the carpal tunnel syndrome: randomised "sham" controlled trial. BMJ. 1998 Mar 7;316(7133):731-5. doi: 10.1136/bmj.316.7133.731. PMID 9529407
- [Background] Totten PA, Hunter JM. Therapeutic techniques to enhance nerve gliding in thoracic outlet syndrome and carpal tunnel syndrome. Hand Clin. 1991 Aug;7(3):505-20. PMID 1939356
- [Background] Page MJ, O'Connor D, Pitt V, Massy-Westropp N. Therapeutic ultrasound for carpal tunnel syndrome. Cochrane Database Syst Rev. 2013 Mar 28;2013(3):CD009601. doi: 10.1002/14651858.CD009601.pub2. PMID 23543580
- [Background] Horng YS, Hsieh SF, Tu YK, Lin MC, Horng YS, Wang JD. The comparative effectiveness of tendon and nerve gliding exercises in patients with carpal tunnel syndrome: a randomized trial. Am J Phys Med Rehabil. 2011 Jun;90(6):435-42. doi: 10.1097/PHM.0b013e318214eaaf. PMID 21430512